CLINICAL TRIAL: NCT03520998
Title: A Prospective, Randomized, Double-Blind, Dose-Comparison Concurrent Control Study to Assess the Safety and Tolerability of GRF6019 Infusions in Subjects With Mild to Moderate Alzheimer's Disease
Brief Title: A Randomized Study to Assess the Safety of GRF6019 Infusions in Subjects With Mild to Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alkahest, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALK6019-201
Record Dates: First submitted 2018-04-25; First posted 2018-05-11 (Actual); Results first posted 2020-11-05 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2018-08

CONDITIONS: Alzheimer Disease; Mild to Moderate Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GRF6019 Low Dose (Experimental): Subjects will receive a low dose of GRF6019 for 5 consecutive days at Week 1 and Week 13.
  Interventions: Drug: GRF6019
- GRF6019 High Dose (Experimental): Subjects will receive a high dose of GRF6019 for 5 consecutive days at Week 1 and Week 13.
  Interventions: Drug: GRF6019

INTERVENTIONS:
Drug: GRF6019 — GRF6019 for IV infusion

SUMMARY:
This study is evaluating the safety, tolerability, and feasibility of GRF6019, a plasma-derived product, administered as an intravenous (IV) infusion, to subjects with mild to moderate Alzheimer's disease.

DETAILED DESCRIPTION:
This is a randomized, double-blind, dose-comparison concurrent control study to assess the safety, tolerability, and feasibility of GRF6019, a plasma-derived product, administered by intravenous (IV) infusion to subjects with mild to moderate Alzheimer's disease.

Subjects will be randomized 1:1 to a low dose or a high dose of active treatment in a double-blind manner. All subjects will receive one infusion per day at the randomized dose for 5 consecutive days during Week 1 and, again, during Week 13 (for a total of 10 doses per subject). All IV infusions will take place at an inpatient research unit while the follow-up visits after each treatment period will be on an outpatient basis. Subjects will participate for a total of 6 months in this study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable AD based upon the National Institute on Aging-Alzheimer's Association (NIA-AA) Criteria
* MMSE Score 12-24 inclusive
* Modified Hachinski Ischemia Scale (MHIS) score of ≤ 4
* Provided a signed and dated informed consent form (either the subject and/or subject's legal representative as well as the trial partner)

Exclusion Criteria:

* Evidence of clinically relevant neurological disorder(s) other than probable AD
* History of blood coagulation disorders or hypercoagulability; any concurrent use of an anticoagulant therapy. (e.g., heparin, warfarin, thrombin inhibitors, Factor Xa inhibitors). Use of antiplatelet drugs (e.g., aspirin or clopidogrel) is acceptable.
* Initiation or change in the dosage of cholinesterase inhibitors (AChEI), memantine, Axona, vitamin E supplementation or selegiline within 3 months prior to screening.
* Heart disease (or history thereof), as evidenced by myocardial infarction, unstable, new onset or severe angina, or congestive heart failure (New York Association Class II, III or IV) in the 6 months prior to dosing; uncontrolled high blood pressure (systolic blood pressure of 160 mmHg or higher and/or diastolic blood
* Prior hypersensitivity reaction to any human blood product or intravenous infusion; any known clinically significant drug allergy.
* Treatment with any human blood product, including transfusions and intravenous immunoglobulin, during the 6 months prior to screening.
* History of immunoglobulin A (IgA), haptoglobulin or C1 inhibitor deficiency; stroke, anaphylaxis, or thromboembolic complications of intravenous immunoglobulins.
* Hemoglobin <10 g/dL in women; and <11 g/dL in men.

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2019-05-24 (Actual); Study Completion 2019-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alkahest Medical Monitor, Study Director — Alkahest, Inc.
Locations (10):
- United States (10):
  - Synergy East, Lemon Grove, California
  - CNS Network, Long Beach, California
  - Pacific Research Network, San Diego, California
  - MD Clinical, Hallandale, Florida
  - Miami Jewish Health Systems, Miami, Florida
  - Behavioral Clinical Research, North Miami, Florida
  - Bioclinica Research, Orlando, Florida
  - Princeton Medical Institute, Princeton, New Jersey
  - Serenity Inpatient, DeSoto, Texas
  - PRA Health Sciences, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- GRF6019 Low Dose: Low dose of GRF6019 for 5 consecutive days at Weeks 1 and 13
- GRF6019 High Dose: High dose of GRF6019 for 5 consecutive days at Weeks 1 and 13
Period: Overall Study
Arm/Group | GRF6019 Low Dose | GRF6019 High Dose
Started | 24 | 23
Completed | 18 | 21
Not Completed | 6 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GRF6019 Low Dose | GRF6019 High Dose | Total
Number analyzed (Participants) | 24 | 23 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.9 (6.26) | 72.7 (7.21) | 74.3 (6.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 29
  Male | 9 | 9 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 7 | 15
  Not Hispanic or Latino | 16 | 16 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 23 | 19 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 23 | 47

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Treatment-emergent Adverse Events (Safety)
Description: Treatment-emergent adverse events identified by MedDRA preferred term and grouped by MedDRA System Organ Class
Time Frame: Baseline to 6 months
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | GRF6019 Low Dose | GRF6019 High Dose
Number analyzed (Participants) | 24 | 23
Participants | 18 | 20

2. Secondary Outcome: The Mini-Mental State Examination (MMSE)
Description: Changes in scores on the MMSE. The MMSE consists of 5 components: orientation to time and place, registration of 3 words, attention and calculation, recall of 3 words, and language. The scores from the 5 components are summed to obtain the overall MMSE total score. The MMSE total score can range from 0 to 30, with higher scores indicating better cognition.
Time Frame: Baseline and 6 months
Population: Evaluable Set and Per Protocol Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GRF6019 Low Dose | GRF6019 High Dose
Number analyzed (Participants) | 21 | 22
score on a scale | -1.0 (4.3) | 1.5 (3.9)

3. Secondary Outcome: Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADASCog/11)
Description: Changes in scores on the 11-item ADASCog/11. The ADAS-Cog/11 includes 11 items assessing cognitive function. The domains include memory, language, praxis, and orientation. There are 70 possible points. Higher scores reflect greater cognitive impairment.
Time Frame: Baseline and 6 months
Population: Evaluable Set and Per Protocol Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GRF6019 Low Dose | GRF6019 High Dose
Number analyzed (Participants) | 21 | 22
score on a scale | -0.4 (5.1) | -0.9 (4.3)

4. Secondary Outcome: The Clinical Dementia Rating Scale - Sum of Boxes (CDR-SOB)
Description: Changes in the CDR-SOB. The CDR characterizes functioning in 6 domains: memory, orientation, judgment and problem solving, community affairs, home and hobbies and personal care. The score is obtained by summing each of the domain box scores. Scores range from 0 to 18 with higher scores reflecting worse cognition.
Time Frame: Baseline and 6 months
Population: Evaluable Set and Per Protocol Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GRF6019 Low Dose | GRF6019 High Dose
Number analyzed (Participants) | 21 | 22
score on a scale | -0.03 (2.3) | 0.21 (1.7)

5. Secondary Outcome: The Alzheimer's Disease Cooperative Study - Activities of Daily Living (ADCS-ADL23)
Description: Changes in the ADCS-ADL23. The ADCS-ADL23 assesses basic and instrumental activities of daily living covering physical and mental functioning and independence in self-care. The score ranges from 0 to 78 with higher scores indicating less functional impairment.
Time Frame: Baseline and 6 months
Population: Evaluable Set and Per Protocol Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GRF6019 Low Dose | GRF6019 High Dose
Number analyzed (Participants) | 21 | 22
score on a scale | -0.7 (7.4) | -1.3 (4.6)

6. Secondary Outcome: The Alzheimer's Disease Cooperative Study - Clinical Global Impression of Change (ADCS-CGIC)
Description: The ADCS-CGIC focuses on clinicians' observations of change in the subject's cognitive, functional, and behavioral performance since the beginning of a trial. The ADCS-CGIC is a 7-point scale with lower values (<4) representing an improvement, higher values (>4) representing a worsening, and a value of 4 indicating no change.
Time Frame: Baseline and 6 months
Population: Evaluable Set and Per Protocol Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GRF6019 Low Dose | GRF6019 High Dose
Number analyzed (Participants) | 21 | 22
score on a scale | 4.1 (0.8) | 4.1 (0.7)

7. Secondary Outcome: The Neuropsychiatric Inventory Questionnaire (NPI-Q)
Description: Change on the NPI-Q. The NPI-Q comprises 12 domains: delusions, hallucinations, dysphoria, apathy, euphoria, disinhibition, aggressivity and restlessness, irritability, anxiety aberrant motor behavior, appetite and eating disorders, and nocturnal behavior. The severity of the reported symptoms is assessed on a 3-point scale. The total severity score can range from 0 to 36 with higher scores representing worse severity.
Time Frame: Baseline and 6 months
Population: Evaluable Set and Per Protocol Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | GRF6019 Low Dose | GRF6019 High Dose
Number analyzed (Participants) | 21 | 22
score on a scale | -2.3 (3.8) | -1.2 (3.1)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | GRF6019 Low Dose | GRF6019 High Dose
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/24 | 2/23
Other Adverse Events (participants affected / at risk) | 12/24 | 14/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GRF6019 Low Dose (N=24) | GRF6019 High Dose (N=23)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GRF6019 Low Dose (N=24) | GRF6019 High Dose (N=23)
Infusion site extravasation (General disorders) | 3 (3) | 2 (2)
Infusion site haematoma (General disorders) | 1 (1) | 4 (4)
Headache (Nervous system disorders) | 3 (4) | 5 (7)
Amylase increased (Investigations) | 1 (1) | 2 (3)
Lipase increased (Investigations) | 1 (1) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-11-02): https://cdn.clinicaltrials.gov/large-docs/98/NCT03520998/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-09): https://cdn.clinicaltrials.gov/large-docs/98/NCT03520998/SAP_001.pdf